CLINICAL TRIAL: NCT03213483
Title: Soft Tissue Augmentation Using Deepithelialized Free Gingival Graft Compared to Connective Tissue Graft in Management of Miller Class I and II Gingival Recession. A Randomized Controlled Clinical Trial
Brief Title: Soft Tissue Augmentation Using Deepithelialized Free Gingival Graft Compared to Connective Tissue Graft in Management of Miller Class I and II Gingival Recession.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Mashaly, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Deepfggvsctg
Record Dates: First submitted 2017-07-06; First posted 2017-07-11 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Gingival Recession
Keywords: gingival recession; connective tissue graft; deepithelialized free gingival graft; free gingival graft
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: Parallel groups, randomized clinical trial
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Single blinded:
  * Blinding of the participants is not applicable.
  * Blinding of the operator is not applicable.
  * Outcome assessor (primary and secondary outcomes) & biostatistician will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subepithelial connective tissue graft (Active Comparator): Patients will receive a coronally advanced flap surgery with a subepithelial connective tissue graft for recession coverage.
  Interventions: Procedure: Coronally advanced flap and subepithelial connective tissue graft
- De-epithelialized free gingival graft (Experimental): Patients will receive a coronally advanced flap surgery with a de-epithelialized free gingival graft for recession coverage.
  Interventions: Procedure: Coronally advanced flap and deepithelialized free gingival graft

INTERVENTIONS:
Procedure: Coronally advanced flap and subepithelial connective tissue graft — The connective tissue graft is obtained by a single line incision from the palate.
  Arms: Subepithelial connective tissue graft
Procedure: Coronally advanced flap and deepithelialized free gingival graft — The connective tissue graft is obtained by deepithelialization of a free gingival graft.
  Arms: De-epithelialized free gingival graft

SUMMARY:
The aim of this study will be to clinically assess the soft tissue augmentation achieved by the de-epithelialized free gingival graft with coronally advanced flap versus the subepithelial connective tissue graft with coronally advanced flap as root coverage procedures for management of patients with Miller class I and II gingival recession.

DETAILED DESCRIPTION:
Evidence from the literature showed that coronally advanced flap was a predictable method for root coverage. The addition of a connective tissue graft was also found to improve the outcome of obtaining complete root coverage in Miller class I and II gingival recession. Many different connective tissue graft-harvesting techniques have been utilized. These techniques aimed at reducing patient morbidity by primary closure of the palatal flap to achieve primary intention wound healing. However, they had the limitation of requiring an adequate thickness of the palatal fibromucosa in order to prevent desquamation of the undermined flap and compromised vasculature.

On the other hand, the free gingival graft surgical technique was also unaccepted esthetically due to the white scar and irregularities produced at the monolingual junction.

Moreover, despite the fact that the free gingival graft had its limitation of being associated with greater post-operative pain, discomfort and bleeding due to healing by secondary intention in 2-4 weeks, nevertheless, this technique was much easier to perform and could be used even in cases of thin palatal fibromucosa.

The evidence in literature comparing patient morbidity and root coverage outcomes between these two techniques is minimal. Studies by Griffin et al. (2006) and Wessel and Tatakis (2008) reported increased incidence of post-operative pain with free gingival grafts. However, a recently study by Zucchelli et al. (2010) compared post-operative morbidity and root coverage outcomes in patients treated with trap-door connective tissue graft and de-epithelialized free gingival graft found no statistically significant differences in pain killer consumption, post-operative discomfort and bleeding between the two groups.

Still very few studies measured the effect of different connective tissue graft harvesting techniques on gingival thickness. And even in the study by Zucchelli et al. (2010), only speculative explanation was given regarding the increase of gingival thickness in case of a de-epithelialized free gingival graft than subepithelial connective tissue graft.

Gingival thickness was proved to be an important factor for the etiology of gingival recession as thick gingival tissues are able to confine the inflammation within the region of the gingival sulcus and prevent its extension to destroy the outer gingival tissue leading to gingival recession.

Therefore, this study will monitor the effect of different connective tissue harvesting techniques (De-epithelialized free gingival graft versus subepithelial connective tissue graft) on gingival thickness enhancement. It will also evaluate the de-epithelialized free gingival graft as a harvesting mechanism for connective tissue graft in terms of patient morbidity and root coverage outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years or older.
2. Periodontally and systemically healthy.
3. Buccal recession defects classified as either Miller class I or II.
4. Presence of identifiable Cementoenamel juction (Zucchelli et al., 2010).
5. Clinical indication and/or patient request for recession coverage.
6. O'Leary index less than 20% (O'Leary et al., 1972).

Exclusion Criteria:

1. Miller class III or IV recession defects.
2. Pregnant females.
3. Smokers as smoking is a contraindication for any plastic periodontal surgery (Khuller, 2009).
4. Handicapped and mentally retarded patients.
5. Patients undergoing radiotherapy.
6. Teeth with cervical restorations, abrasion.
7. Presence of systemic disease that would affect wound healing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2019-05-27 (Actual); Study Completion 2019-07-27 (Actual)

PRIMARY OUTCOMES:
Gingival Thickness | 6 months
  Thickness of the gingival tissues 2 mm from the free gingival margin

SECONDARY OUTCOMES:
Percentage of root coverage | 6 months
  (Preoperative vertical recession - Postoperative vertical recession/preoperative vertical recession) x 100.
Root coverage esthetic score | 6 months
  A system proposed for evaluating esthetic outcomes of root coverage procedures.
Post-Operative Pain | Two weeks
  Visual Analogue Scale (VAS) with numbers from 0 to 10 ('no pain' to 'worst pain imaginable') measured daily for the first 2 weeks postoperatively
Post-operative stress | Two weeks
  level of stress experienced by the patients of jeopardizing the palatal wound during the time of healing
Post-operative bleeding | Two weeks
  prolonged hemorrhaging during the post-surgical week reported by the patients measured by a questionnaire as a categorical yes or no question.
Post-operative inability to chew | Two weeks
  Will be described as the level of variation of the patient's eating habits due to the presence of the palatal wound.
Post-Surgical Patient Satisfaction | 6 months
  A 3-item questionnaire is asked and the patients shall use a 7-point answer scale.

CONTACTS AND LOCATIONS:
Overall Officials: Azza Ezz Elarab, Phd, Study Chair — Professor; Noha Ghallab, Phd, Study Director — Professor; Weam El Battawy, Phd, Study Director — Lecturer
Locations (1):
- Faculty of Oral and Dental Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zucchelli G, Mele M, Stefanini M, Mazzotti C, Marzadori M, Montebugnoli L, de Sanctis M. Patient morbidity and root coverage outcome after subepithelial connective tissue and de-epithelialized grafts: a comparative randomized-controlled clinical trial. J Clin Periodontol. 2010 Aug 1;37(8):728-38. doi: 10.1111/j.1600-051X.2010.01550.x. Epub 2010 Jun 24. PMID 20590963